CLINICAL TRIAL: NCT02299986
Title: An InnovaTive Approach to Ventilator-Induced Diaphragmatic Dysfunction
Acronym: ITAVIDD
Status: Completed | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Tom Schepens, MD, MD, University Hospital, Antwerp
Other Study IDs: EC 13/12/131; B300201317057 (Other: Belgian Federal Agency for Medicines and Health products)
Record Dates: First submitted 2014-11-10; First posted 2014-11-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Ventilator-induced Diaphragm Dysfunction; VIDD

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single arm Ultrasound measurement: Ultrasound measurement
  Interventions: Other: Ultrasound measurement

INTERVENTIONS:
Other: Ultrasound measurement — Thickness measurement through ultrasound. The investigators will perform daily ultrasound measurements to assess the evolution in thickness during mechanical ventilation

SUMMARY:
'Ventilator-Induced Diaphragmatic Dysfunction (VIDD) was originally described by Vassilakopoulos and Petrof in 1998, where it is used to cover the effects of mechanical ventilation and respiratory muscle unloading on the diaphragm. A recent article by Grosu and colleagues has demonstrated that the thickness of the diaphragm decreases with about 6% a day in a small cohort of mechanically ventilated patients. This is a longitudinal, single-centre, observational cohort study to examine the long-term effects of invasive mechanical ventilation on the diaphragm, and to study the risk factors associated with VIDD.

ELIGIBILITY:
Inclusion Criteria:

* The patient must suffer from respiratory insufficiency requiring mechanical ventilation

Exclusion Criteria:

* The patient has been hospitalized and mechanically ventilated (invasive or non- invasive) in the period up to 1 year before start of the study.
* The patient is known or suspected to have an anatomical malformation of the diaphragm.
* The patient suffers from a disease that may impair diaphragmatic function:

  * Central neural disease at the level of the brain (Multiple sclerosis, stroke, Arnold-Chiari malformation) and spinal cord (quadriplegia, amyotrophic lateral sclerosis, poliomyelitis, spinal muscular atrophy, syringomyelia).
  * Neural disease of the phrenic nerve (Guillain-Barré syndrome, tumor compression, neuralgic neuropathy, chronic inflammatory demyelinating polyneuropathy, Charcot-Marie-Tooth disease).
  * Disorders of the neuromuscular junction (Myasthenia gravis, Lambert- Eaton syndrome, botulism, organophosphate poisoning).
  * Muscular diseases (muscular dystrophies, myositis (infectious, inflammatory, metabolic).
* The patient is known or suspected to have a psychiatric illness inhibiting his/her cooperation with the study protocol or possibly obscuring the obtained results.
* The patient has been mechanically ventilated for over 24 hours before the first ultrasonographic measurement can be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that are admitted in ICU and who require mechanical ventilation will be screened for inclusion, and participants will be enrolled after informed consent. The study population will be a mixed medical/surgical cohort, selected with non-probability sampling because of the different eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2013-04; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in diaphragm thickness | Participants will be followed during their ICU stay, an expected average of 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Tom Schepens, MD, Principal Investigator — University Hospital, Antwerp
Locations (1):
- Antwerp University Hospital, Edegem, Antwerp, Belgium

REFERENCES:
- [Background] Grosu HB, Lee YI, Lee J, Eden E, Eikermann M, Rose KM. Diaphragm muscle thinning in patients who are mechanically ventilated. Chest. 2012 Dec;142(6):1455-1460. doi: 10.1378/chest.11-1638. PMID 23364680
- [Derived] Schepens T, Verbrugghe W, Dams K, Corthouts B, Parizel PM, Jorens PG. The course of diaphragm atrophy in ventilated patients assessed with ultrasound: a longitudinal cohort study. Crit Care. 2015 Dec 7;19:422. doi: 10.1186/s13054-015-1141-0. PMID 26639081